CLINICAL TRIAL: NCT02654756
Title: Risk of Chronic Kidney Disease Progression
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 13311
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease
Keywords: Risk Assessment
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
While there are proven therapies that slow CKD progression, these therapies can at times be harmful and costly. The ability to accurately predict the risk of CKD progression to ESRD would be extremely valuable. The short term versus lifetime risk of CKD progression should be taken into account when making risk based clinical decisions. In a representative CKD practice, the investigators compared the short term and lifetime risk assessment in our stage 3 CKD patients to determine whether decisions based on a short term risk assessment would underestimate the lifetime risk of CKD progression. The investigators also applied the short term risk assessment to our stage 4 CKD patients to determine the frequency with which ESRD risk may be overestimated in CKD stage 4.

DETAILED DESCRIPTION:
In the US, more than 20 million adults have Chronic Kidney Disease (CKD) and are therefore at increased risk for cardiovascular disease (CVD) and progression to end-stage renal disease (ESRD) as compared to those without CKD. While there have been many substantiated therapies that slow the progression of CKD and improve overall outcomes, clinical decision making is difficult due to the variability of progression of CKD and increased risk of cardiovascular mortality. As these therapies can at times be harmful and costly, the ability to accurately predict the risk of CKD progression would be extremely valuable. Kidney Disease: Improving Global Outcomes (KDIGO) recently incorporated a risk scale that was a reflection of a composite of 5 CKD outcomes: all-cause mortality, CVD mortality, ESRD, acute kidney injury (AKI) and progression of CKD. It is in its infancy and guidelines reflecting this risk stratification have yet to be determined. Several risk prediction tools that have been validated in specific CKD populations but none have been widely accepted and implemented in the clinical setting. These tools incorporate multiple risk factors as compared to the KDIGO risk categories which uses eGFR and urine albumin to creatinine ratio (ACR) to determine the risk of the above mention composite. The KDIGO scale does not take age into account and this may have a major effect on risk stratification. One risk assessment tool that does take the patients' age into account is the risk equation developed from the paper by Tangri N et al. (JAMA 2011;305(15):1553-1559). This equation uses age, sex, serum calcium levels, serum phosphate levels, serum albumin levels and serum bicarbonate levels in addition to GFR and UCR to calculate the risk of progression to ESRD requiring dialysis or transplantation. This risk calculator reflects short term risk as it supplies a 2yr and 5yr progression risk for CKD stage 3 and 4 patients. A Lifetime risk estimator (adjusted for competing risk of death) that uses age, sex and eGFR to define an age and sex specific 10, 20, 30, 40 and lifetime risk for CKD progression was provided by a study by Turin TC et al (J Am Soc Nephrol 2012;23(9):1569-1578). The purpose of this study is to examine the effect of using the 2yr, 5yr and lifetime risk assessment tools on a population of individuals with stage 3 and 4 CKD.

ELIGIBILITY:
Inclusion Criteria:

* Evaluation at least once by a nephrologist in the past year.
* Subjects must have recent pertinent laboratory data within the last 2 years.
* 2 documented creatinine values separated by at least 3 months

Exclusion Criteria:

* Deceased patients
* estimated GFR < 15ml/min
* Patients with Acute Renal Failure (ARF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nephrology outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 623 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Percentage difference in risk levels when comparing short term risk and lifetime risk in patients with CKD stage 3. | 2 to 5 years
Percentage of patients with CKD stage 4 in low, intermediate and high risk categories after assessing short term risk in patients with CKD stage 4. | 2 to 5 years

SECONDARY OUTCOMES:
Assessment ESRD outcomes after risk stratification. | 2 to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Candace Grant, MD, Principal Investigator — NYU Winthrop
Locations (1):
- NYU Winthrop, Mineola, New York, United States